CLINICAL TRIAL: NCT00068614
Title: A Phase I Trial Evaluating The Safety Of Intramuscular Injections Of HER-2 Protein AUTOVAC (PX104.1.6) In Patients With Breast Cancer
Brief Title: HER-2 Protein Vaccine in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PMXA1103; CWRU-030339; CDR0000327784 (Registry Identifier: PDQ (Physician Data Query)); PHARMEXA-PX104.1.6-101
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of HER-2 protein vaccine in treating women who have breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of HER-2 protein AutoVac™ in women with breast cancer.

Secondary

* Determine the ability of this drug to bypass the tolerance to the HER-2 self-protein by raising HER-2 antibodies in these patients.
* Determine the kinetics of the immune response to HER-2/neu in patients treated with this drug.

OUTLINE: This is an open-label, multicenter study.

Patients receive HER-2 protein AutoVac™ intramuscularly at weeks 0, 2, 6, and 10 in the absence of unacceptable toxicity.

Patients are followed for up to 6 weeks.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast, meeting criteria for 1 of the following:

  * Metastatic disease currently in complete or partial response or stable disease

    * Have been receiving a stable endocrine therapy regimen (e.g., aromatase inhibitor, tamoxifen, fulvestrant, or gonadotropin-releasing hormone agonist) for at least 30 days OR status post oophorectomy
  * Completed a course of local and adjuvant systemic therapy for high-risk stage II or III disease (i.e., anticipated 5-year relative survival is no greater than 50%) meeting any of the following staging criteria:

    * Stage IIB with involvement of at least 4 nodes
    * Stage IIIA (T3 disease with involvement of at least 4 nodes)
    * Any stage IIIB or IIIC disease
  * Stage IV with no evidence of disease (e.g., prior resection of local chest wall recurrence with no evidence of disease elsewhere)
* 1+, 2+, or 3+ HER2/neu expression by immunohistochemistry
* Treatment with trastuzumab (Herceptin®) not clinically indicated
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* Absolute neutrophil count at least 1,500/mm^3

Hepatic

* ALT or AST no greater than 2.5 times upper limit of normal (ULN) (5 times ULN for patients with liver metastases)
* Bilirubin no greater than 2 mg/dL (unless due to Gilbert's disease)

Renal

* Creatinine no greater than 2 mg/dL

Cardiovascular

* No history of significant cardiovascular disease
* No myocardial infarction within the past 6 months
* No poorly controlled cardiac arrhythmia
* No New York Heart Association class III or IV heart disease
* LVEF at least 50% by MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy except basal cell skin cancer or adequately treated carcinoma in situ of the cervix
* No concurrent severe autoimmune disease
* No other clinically significant or serious medical disease that would preclude study participation or compromise patient safety or the results of this study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 months since prior trastuzumab
* No prior anticancer vaccine therapy
* No concurrent trastuzumab
* No concurrent immunomodulators (e.g., thalidomide or interferons/interleukins)

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No concurrent low-dose methotrexate or cyclophosphamide
* No concurrent cytotoxic chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent corticosteroids

  * Topical or inhaled steroids are allowed
* No changes to current endocrine therapy regimen (e.g., discontinuation or addition of an agent)

Radiotherapy

* More than 3 months since prior radiotherapy involving more than 25% of the bone marrow
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* No prior bilateral breast procedures

Other

* More than 4 weeks since prior immunosuppressive therapy
* More than 30 days since prior investigational agents or clinical trial participation
* No other concurrent experimental or investigational agents
* No concurrent cyclosporine
* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Overmoyer, MD, FACP, Study Chair — Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center, Cleveland, Ohio, United States